CLINICAL TRIAL: NCT06947317
Title: Relevance of Osteochondral Lesions in Ankle Microinstability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAUL FIGA BARRIOS (Other)
Responsible Party: Sponsor-Investigator, RAUL FIGA BARRIOS, Consultant in the Foot and Ankle Unit of the Department of Orthopedic Surgery and Traumatology, Consorci Sanitari de Terrassa
Organization: Consorci Sanitari de Terrassa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-20-105-055; MED-2022-05 (Other: Universitat Internacional de Catalunya)
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lateral Ligament, Ankle; Cartilage, Articular
Keywords: Cartilage, Articular; Lateral Ligament, Ankle; Arthroscopy; Ankle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REC (Reconstruction Only) Group (Active Comparator): This group underwent only the anterior talofibular ligament (ATFL) repair using the all-inside arthroscopic technique.
  Interventions: Procedure: Arthroscopic anterior talofibular ligament repair
- REC+MIC (Reconstruction with Microfracture) Group (Experimental): This group underwent both the ATFL repair and the additional procedure of curettage and microfracture for the osteochondral lesion of the talus via arthroscopy.
  Interventions: Procedure: Arthroscopic anterior talofibular ligament repair; Procedure: Talar chondral lesion treatment using microfracture technique

INTERVENTIONS:
Procedure: Arthroscopic anterior talofibular ligament repair — This intervention involves an isolated all-inside arthroscopic repair of the anterior talofibular ligament (ATFL) without addressing the coexisting osteochondral lesion of the talus. It is intended for patients with chronic ankle instability and a concomitant talar osteochondral lesion, where only the ligamentous injury is treated. Patients follow a standard rehabilitation protocol with return to sports allowed after 3 months.
Procedure: Talar chondral lesion treatment using microfracture technique — This intervention consists of an arthroscopic debridement and microfracture of a symptomatic osteochondral lesion of the talus. Postoperative rehabilitation is extended due to the cartilage procedure, delaying return to sports until 4 months.
  Arms: REC+MIC (Reconstruction with Microfracture) Group

SUMMARY:
The goal of this clinical trial is to learn if treating only the anterior talofibular ligament (ATFL) tear with ligament repair is as effective as treating both the ligament tear and the associated osteochondral lesion of the talus at the same time in adults with ankle instability and pain.

The main questions it aims to answer are:

* Do patients who undergo both ligament repair and treatment of the cartilage lesion have better clinical and functional outcomes than those who only have the ligament repaired?
* Is there a difference in pain relief, recovery time, and return to physical activity between the two approaches?

Researchers will compare patients who receive isolated ligament repair to those who receive ligament repair plus microfracture surgery to see if treating both injuries provides better results.

Participants will:

* Be randomly assigned to one of the two treatment groups.
* Undergo surgery by the same surgeon.
* Complete questionnaires about ankle function and pain before surgery and at multiple follow-up points.
* Have physical exams and imaging to assess ankle stability and healing.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the clinical relevance of concomitant osteochondral lesions of the talus in patients undergoing surgical treatment for chronic ankle instability (CAI). Despite successful ligament reconstruction, a substantial proportion of patients report persistent pain, possibly due to associated intra-articular pathology. The study aims to determine whether addressing the osteochondral lesion during the same surgical procedure provides additional clinical or functional benefit compared to isolated ligament repair.

Sixty adult patients with symptomatic CAI and a concomitant talar osteochondral lesion (≤150 mm², Berndt-Harty stage I-IIb) were randomly assigned to two parallel groups. Both groups underwent arthroscopic all-inside anterior talofibular ligament (ATFL) repair. In the experimental group, additional curettage and microfracture of the osteochondral lesion were performed. A standardized rehabilitation protocol was followed, with return to sport permitted at three months for the isolated repair group, and four months for the combined intervention group due to the more extensive surgical gesture.

Primary and secondary outcomes were assessed using validated scales (AOFAS, Karlsson, SEFAS, and VAS) at baseline, and at 1, 3, 6, 12, and 24 months postoperatively. The minimum follow-up period was two years. Statistical analysis included mixed ANOVA for repeated measures and adjustment for multiple comparisons. The study was powered to detect clinically significant differences in AOFAS scores between groups, with a sample size of 30 per group allowing for 20% attrition.

This study addresses a current gap in the literature regarding the management of osteochondral lesions in CAI and provides level I evidence to guide treatment decisions in patients with combined ligamentous and chondral pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an anterior talofibular ligament (ATFL) tear
* Presence of an osteochondral lesion (OCL) <150 mm²
* OCL classified as stage I-IIb according to the Berndt & Harty classification
* Clinical signs of ankle instability
* Pain in the tibiotalar joint
* Incomplete symptom resolution after prior non-surgical treatment
* Age over 18 years

Exclusion Criteria:

* Congenital or post-traumatic bone deformity of the ankle or foot on the affected side
* Previous surgery on the affected limb
* Neuromuscular disorders
* Generalized joint hyperlaxity (Beighton Score)
* Medial ankle instability (due to deltoid ligament injury)
* Presence of OCL >150 mm²
* Presence of multiple OCLs or other concomitant intra- or extra-articular lesions
* History of ankle fracture
* Lack of signed informed consent
* Body mass index >30 Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Change in AOFAS (American Orthopaedic Foot and Ankle Society) score | Baseline, 3 months, 6 months, 12 months, and 24 months postoperative
  Evaluation of functional outcome using the AOFAS Ankle-Hindfoot Scale, which combines pain, function, and alignment. The AOFAS score ranges from 0 (severe disability) to 100 (normal function).

SECONDARY OUTCOMES:
Change in Karlsson score | Baseline, 3 months, 6 months, 12 months, and 24 months postoperative
  Assessment of ankle instability and function using the Karlsson scoring scale. The Karlsson score ranges from 0 (severe instability and dysfunction) to 100 (normal ankle function).
Change in SEFAS (Self-reported Foot and Ankle Score) | Baseline, 3 months, 6 months, 12 months, and 24 months postoperative
  Patient-reported questionnaire evaluating pain and function in the foot and ankle. The SEFAS score ranges from 0 (severe disability) to 48 (normal function).
Change in Visual Analogue Scale (VAS) for pain | Baseline, 1 month, 3 months, 6 months, 12 months, and 24 months postoperative
  Patient-reported level of pain using a 10-point visual scale. The Visual Analogue Scale (VAS) for pain ranges from 0 (no pain) to 10 (worst imaginable pain).
Surgical failure and reintervention rate | Any time during the 24-month follow-up period
  Number of participants requiring additional surgical procedures on the same ankle due to persistent symptoms or complications related to the initial intervention.

CONTACTS AND LOCATIONS:
Overall Officials: RAÚL FIGA BARRIOS, Principal Investigator — Consultant in the Foot and Ankle Unit of the Department of Orthopedic Surgery and Traumatology
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Spain, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article will be made available upon reasonable request to the corresponding author, for purposes of academic and non-commercial research. Requesters will need to provide a methodologically sound proposal and agree to a data access agreement to ensure confidentiality and appropriate use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 6 months after publication of the primary results and will remain available for a period of 5 years.
Access Criteria: De-identified individual participant data (IPD) that underlie the results reported in this article will be made available upon reasonable request to the corresponding author, for purposes of academic and non-commercial research. Requesters will need to provide a methodologically sound proposal and agree to a data access agreement to ensure confidentiality and appropriate use.

REFERENCES:
- [Derived] Figa Barrios R, Mora-Guix JM, Roza Miguel PO, Vila-Rico J. Additional cartilage treatment for small defects in chronic ankle instability shows no mid-term benefit and delays recovery: a randomized controlled trial. J Orthop Traumatol. 2025 Oct 9;26(1):67. doi: 10.1186/s10195-025-00880-9. PMID 41065921